CLINICAL TRIAL: NCT03902080
Title: A Phase 3 Double-Blind, Randomized, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy, Safety and Tolerability of Vibegron in Men With Overactive Bladder (OAB) Symptoms on Pharmacological Therapy for Benign Prostatic Hyperplasia (BPH)
Brief Title: Study to Evaluate the Efficacy, Safety and Tolerability of Vibegron in Men With Overactive Bladder (OAB) Symptoms on Pharmacological Therapy for Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Urovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URO-901-3005; 2018-003135-30 (EudraCT Number)
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-06

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Benign Prostatic Hyperplasia; Vibegron; Beta-3 adrenergic receptor (ß3-AR); ß3-AR agonist
MeSH Terms: conditions — Urinary Bladder, Overactive; Prostatic Hyperplasia | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vibegron 75 mg (Experimental): Participants will receive vibegron 75 milligrams (mg) orally once daily for 24 weeks.
  Interventions: Drug: Vibegron
- Placebo (Placebo Comparator): Participants will receive matching placebo orally once daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vibegron — oral administration
  Other Names: RVT-901; MK-4618; KRP-114V; URO-901
  Arms: Vibegron 75 mg
Drug: Placebo — oral administration
  Arms: Placebo

SUMMARY:
This study will assess the efficacy of vibegron compared with placebo in men with overactive bladder (OAB) symptoms on pharmacological therapy for benign prostatic hyperplasia (BPH) as defined by micturition and urgency episodes.

ELIGIBILITY:
Inclusion Criteria:

* Participant should have been on and agree to continue to stay on a stable dose of benign prostatic hyperplasia (BPH) treatment with either a) alpha blocker monotherapy or b) alpha blocker + 5 alpha reductase inhibitor.
* Participant has an International Prostate Symptom Score total score of ≥ 8
* Participant has a prostate-specific antigen level < 4 nanograms per milliliter (ng/mL), or if ≥ 4 ng/mL but ≤ 10 ng/mL, prostate cancer has been ruled out to the satisfaction of the investigator
* Participant must have both additional qualifications based on the 3-day Bladder Diary period: a) having an average of ≥ 8 but ≤ 20 micturition episodes per day over the 3-day diary period, and (b) having an average of ≥ 3 urgency episodes per day over the 3-day diary period
* Participant must have a post void residual volume value of < 100 mL
* Having at least 2 average nocturia episodes per night based on 3-day Bladder Diary at baseline. Nocturia is defined as waking to pass urine during the main sleep period.

Exclusion Criteria:

* Participant has a history of 24-hour urine volume greater than 3,000 mL
* Has lower urinary tract pathology that could, in the opinion of the investigator, be responsible for urgency, frequency, or incontinence
* Has a history of prostate surgery, including minimally invasive transurethral or transrectal procedures, procedural treatments for BPH within 6 months of Screening or has a planned prostate surgery
* Has a history of urinary retention requiring an intervention (e.g., catheterization) for any reason
* Has maximum urinary flow (Qmax) < 5.0 mL/second with a minimum voided volume of 125 mL
* Has a history of or current nocturnal polyuria
* Has an active or recurrent (> 3 episodes per year) urinary tract infection by clinical symptoms or laboratory criteria (≥ 5 white blood cells/high power field [hpf] with presence of red blood cell [RBC] and/or a positive urine culture, defined as ≥ 10^5 colony forming units (CFU)/mL (i.e., 100 × 10^3 CFU/mL in a single specimen)
* Has uncontrolled hyperglycemia (defined as fasting blood glucose > 150 milligrams per deciliter (mg/dL) or 8.33 millimoles per liter (mmol/L) or non-fasting blood glucose > 200 mg/dL or 11.1 mmol/L) or, if in the opinion of the investigator, is uncontrolled
* Has uncontrolled hypertension (systolic blood pressure of ≥ 180 millimeters of mercury (mmHg) and/or diastolic blood pressure of ≥ 100 mmHg) or has a resting heart rate (by pulse) > 100 beats per minute (min)
* Has a history of cerebral vascular accident, transient ischemic attack, unstable angina, myocardial infarction, coronary artery interventions (e.g., coronary artery bypass grafting or percutaneous coronary interventions [e.g., angioplasty, stent insertion]), or neurovascular interventions (e.g., carotid artery stenting) within 6 months prior to the Screening Visit
* Has alanine aminotransferase or aspartate aminotransferase > 2.0 times the upper limit of normal (ULN), or bilirubin (total bilirubin) > 1.5 × ULN (or > 2.0 × ULN if secondary to Gilbert syndrome or pattern consistent with Gilbert syndrome)
* Has an estimated glomerular filtration rate < 30 mL/min/1.73 meters squared (m^2)
* Has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstances that might, in the opinion of the investigator, confound the results of the study, interfere with the participant's ability to comply with the study procedure, or make participation in the study not in the participant's best interest

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1105 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Urovant Sciences
Locations (140):
- United States (75):
  - Urology Centers of Alabama, Homewood, Alabama
  - Private Practice, Huntsville, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Gen1 Research- Arizona Urology Specialists, Glendale, Arizona
  - Urological Associates Of Southern Arizona, Tucson, Arizona
  - California Research Medical Group, Inc., Fullerton, California
  - San Diego Clinical Trials, La Mesa, California
  - Clinical Trials Research, Lincoln, California
  - West Coast Urology, Los Alamitos, California
  - American Institute of Research, Los Angeles, California
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - Northern California Research Corp, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - Urology Specialists of Southern California (USSC), Sherman Oaks, California
  - Skyline Urology, Torrance, California
  - Urology Associates - Urology, Denver, Colorado
  - Imagine Research of Palm Beach County - Urology, Boynton Beach, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Urological Research Network Corp, Hialeah, Florida
  - LCC Medical Research Institute, Miami, Florida
  - Quantum Clinical Trials, Miami, Florida
  - Private Practice, Orlando, Florida
  - Urology Center Of Florida, Pompano Beach, Florida
  - Pinellas Urology, Inc., St. Petersburg, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Florida Urology Partners, LLP, Tampa, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Meridian Clinical Research - Urology, Savannah, Georgia
  - Idaho Urologic Institute, Meridian, Idaho
  - NorthShore University Health System, Glenview, Illinois
  - First Urology, Jeffersonville, Indiana
  - The Iowa Clinic, West Des Moines, Iowa
  - GU Research Network/Wichita Urology Group, Wichita, Kansas
  - DelRicht Research, New Orleans, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Boston Clinical Trials Inc - Urology, Boston, Massachusetts
  - Mens Health Boston - Urology, Chestnut Hill, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Beaumont Hospital Royal Oak - Urology Research, Royal Oak, Michigan
  - CentraCare Clinic - Adult & Pediatric Urology, Sartell, Minnesota
  - Poplar Bluff Urology, Poplar Bluff, Missouri
  - Adult & Pediatric Urology P.C. - Urology, Omaha, Nebraska
  - Excel Clinical Research - Internal Medicine, Las Vegas, Nevada
  - Private Practice, Las Vegas, Nevada
  - Premier Urology Group, LLC, Edison, New Jersey
  - New Jersey Urology NJU, Englewood, New Jersey
  - New Jersey Urology, LLC, Mount Laurel, New Jersey
  - New Jersey Urology, LLC, Voorhees Township, New Jersey
  - Albany Medical College, Albany, New York
  - Western New York Urology Associates, Buffalo, New York
  - AccuMed research Asociates, Garden City, New York
  - Urological Surgeons of Long Island, Garden City, New York
  - Manhattan Research Associates, New York, New York
  - Columbia University Medical Center - Clinical Research, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Advanced Urology Centers of NY, A Division of Integrated Medical Professionals (IMP), Plainview, New York
  - Private Practice, Poughkeepsie, New York
  - Duke Medical Center - Urology, Durham, North Carolina
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Alliance Urology Specialists - Greensboro, Greensboro, North Carolina
  - Triad Clinical Trials, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Associated Urologists of North Carolina - Urology, Raleigh, North Carolina
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Lowcountry Urology, North Charleston, South Carolina
  - Urology Clinics of North Texas, Dallas, Texas
  - Advances In Health, Inc., Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - Discovery Clinical Trials, San Antonio, Texas
  - Baylor Scott & White Medical Center, Temple, Texas
  - Wasatch Clinical Research LLC, Salt Lake City, Utah
  - Urology of Virginia (UVA), Virginia Beach, Virginia
  - Seattle Urology Research Center, Burien, Washington
- Belgium (7):
  - Uz Antwerpen, Edegem, Antwerpen
  - Algemeen Stedelijk Ziekenhuis, Aalst, Oost-Vlaanderen
  - Onze-Lieve-Vrouwziekenhuis VZW - Campus Aalst, Aalst, Oost-Vlaanderen
  - AZ Maria Middelares - Campus Maria Middelares, Ghent, Oost-Vlaanderen
  - UZ Leuven - Campus Gasthuisberg, Leuven, Vlaams Brabant
  - AZ Delta - Campus Wilgenstraat, Roeselare, West-Vlaanderen
  - CHU de Liège - Domaine Universitaire du Sart Tilman - Urologie, Liège
- Canada (8):
  - Private Practice, Brampton, Ontario
  - Bluewater Clinical Research Group Inc, Sarnia, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Diex Research Quebec Inc., Québec, Quebec
  - Centre Hospitalier Universitaire De Sherbrooke (CHUS), Sherbrooke, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
  - Diex Research Victoriaville Inc., Victoriaville, Quebec
- Hungary (8):
  - University of Szeged, Szeged, Csongrád megye
  - DRC Kft., Sopron, Győr-Moson-Sopron
  - Semmelweis Egyetem, Budapest
  - Jahn Ferenc Dél-Pesti Kórház és Rendelointézet, Budapest
  - Szarka Ödön Egyesitett Egeszsegügyi es Szocialis Intezmeny, Csongrád
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókór, Nyíregyháza
  - Uro-Clin Kft., Pècs
  - Szent Borbala Korhaz, Tatabánya
- Lithuania (10):
  - Kaunas Hospital of Lithuanian Universoity of Health Sciences, Kaunas, Kaunas County
  - JSC Saules seimos medicinos centras, Kaunas, Kaunas County
  - Uab "Vakk", Kaunas, Kaunas County
  - Hospital of University of Health Sciences Kauno Klinikos, Kaunas, Kaunas County
  - Respublikine Klaipedos ligonine - Urology, Klaipėda, Klaipėda County
  - Klaipedos Universitetine Ligonine (Klaipeda Hospital), Klaipėda, Klaipėda County
  - National Cancer Institute, Vilnius, Vilnius County
  - Republican Vilnius University Hospital, Vilnius, Vilnius County
  - Vilnius University Hospital Santariskiu Klinikos, Vilnius, Vilnius County
  - Vilnius City Clinical Hospital, Vilnius, Vilnius County
- Poland (13):
  - EuroMediCare Szpital Specjalistyczny z Przychodnia, Wroclaw, Dolnoslaskie Województwo
  - Clinical Research Center Sp. z o.o., Medic-R Sp. K., Poznan, Greater Poland Voivodeship
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Wojewodzki Szpital Specjalist, Wroclaw, Lower Silesian Voivodeship
  - NZOZ Specjalista, Kutno, Lódzkie
  - ETG Lodz, Lodz, Lódzkie
  - Centrum Medyczne PROMED, Krakow, Malopolskie Województwo
  - Szpital Specjalistyczny Slupsk, Słupsk, Pomeranian Voivodeship
  - Centrum Urologiczne sp. z o.o., Mysłowice, Silesian Voivodeship
  - Centrum Medyczne Linden, Krakow
  - Medicome Sp. z o.o., Oświęcim
  - Nzoz Heureka, Piaseczno
  - Lexmedica Hanna Durbajlo-Gradziel, Wroclaw
- Portugal (6):
  - Hospital Garcia de Orta, Almada
  - Centro Clínico Académico Braga, Hospital de Braga, Braga
  - Hospital Senhora de Oliveiro Guimaraes EPE, Guimarães
  - H. Egas Moniz. Centro Hospitalar Lisboa Ocidental, Lisbon
  - Hospital de Santa Maria, Lisbon
  - H. Santo António. Centro Hospitalar do Porto, Porto
- Spain (13):
  - Hospital Santiago Apostol, Miranda de Ebro, Burgos
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Hospital General Universitario Gregorio Marañón, Majadahonda, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital del Mar, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Clínica Universitaria de Navarra, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - H.U. Virgen de la Victoria, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Urovant is committed to sharing patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Data requests will be reviewed and approved on the basis of scientific merit. All data provided will be anonymized according to applicable laws and regulations.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be made available within 24 months after study completion and will be accessible for a time frame appropriate for the approved proposal.
Access Criteria: Access to these clinical trial data can be requested by emailing medinfo@urovant.com and will be provided following Urovant review and approval of a research proposal and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Rovner ES, Owens-Grillo J, Thomas E, Herschorn S, Peters KM, Staskin D, Mujais S. Bladder Function and Safety of Vibegron in Men With Overactive Bladder Receiving Treatment for Benign Prostatic Hyperplasia: Outcomes From the Phase 3 Randomized Controlled COURAGE Trial. Neurourol Urodyn. 2026 Feb;45(2):299-304. doi: 10.1002/nau.70199. Epub 2025 Dec 9. PMID 41363221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 3, randomized, double-blind, placebo-controlled, 2 part, parallel-group, multicenter study to evaluate the safety, tolerability, and efficacy of vibegron in men with symptoms of overactive bladder (OAB) on stable doses of pharmacological therapy for benign prostatic hyperplasia (BPH).
Pre-assignment Details: Participants were enrolled in 82 sites across 8 countries. One randomized participant enrolled in the placebo group did not receive double-blind medication.
Groups:
- Vibegron 75 Milligrams (mg) Once Daily (QD): Participants were randomized 1:1 to receive 75 mg of Vibegron tablet orally QD
- Placebo: Participants were randomized 1:1 to receive matching placebo tablet orally QD
Period: Overall Study
Arm/Group | Vibegron 75 Milligrams (mg) Once Daily (QD) | Placebo
Started | 551 | 554
Received at Least 1 Dose of Double-blind Medication | 551 | 553
Completed | 484 | 481
Not Completed | 67 | 73
Not completed — Adverse Event | 17 | 15
Not completed — Withdrawal by Subject | 28 | 35
Not completed — Lost to Follow-up | 6 | 7
Not completed — Other | 3 | 5
Not completed — Non compliance | 4 | 3
Not completed — Physician Decision | 5 | 1
Not completed — Protocol Violation | 3 | 3
Not completed — Lack of Efficacy | 1 | 3
Not completed — Withdrawn prior to dosing | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set consists of all randomized participants who took at least 1 dose of double-blind study treatment and had at least 1 evaluable change from Baseline mictruition
Groups:
- Total: Total of all reporting groups
Arm/Group | Vibegron 75 Milligrams (mg) Once Daily (QD) | Placebo | Total
Number analyzed (Participants) | 538 | 542 | 1080
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (8.06) | 67.4 (7.92) | 67.1 (7.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 538 | 542 | 1080
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 14 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 58 | 48 | 106
  White | 471 | 475 | 946
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 12 in the Average Number of Micturition Episodes Per Day
Description: Micturition was defined as the number of times a participant voided in the toilet as indicated on the Bladder Diary. Baseline was defined as the last non-missing result on or prior to the randomization date. Change from baseline was calculated as the post-baseline value minus the baseline value. Daily Averages were calculated as the sum of the event type on Complete Diary Days divided by the number of Complete Diary Days.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only those participants with data available at specified time points have been presented.
Measure: Least Squares Mean (Standard Error); unit: Micturitions per day
Arm/Group | Vibegron 75 Milligrams (mg) Once Daily (QD) | Placebo
Number analyzed (Participants) | 503 | 507
Micturitions per day | -2.04 (0.109) | -1.30 (0.109)
Statistical Analysis 1: Comparison: Vibegron 75 Milligrams (mg) Once Daily (QD) vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least square mean difference = -0.74, 95% CI 2-sided [-1.02 to -0.46], Standard Error of Mean 0.142

2. Primary Outcome: Change From Baseline at Week 12 in the Average Number of Urgency Episodes (Need to Urinate Immediately) Per Day
Description: Urgency was defined as the number of times a participant checked that they had the need to urinate immediately as indicated on the Bladder Diary. Baseline was defined as the last non-missing result on or prior to the randomization date. Change from baseline was calculated as the post-baseline value minus the baseline value. Daily Averages were calculated as the sum of the event type on Complete Diary Days divided by the number of Complete Diary Days.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only those participants with data available at specified time points have been presented.
Measure: Least Squares Mean (Standard Error); unit: Urgency Episodes per Day
Arm/Group | Vibegron 75 Milligrams (mg) Once Daily (QD) | Placebo
Number analyzed (Participants) | 503 | 507
Urgency Episodes per Day | -2.88 (0.164) | -1.93 (0.164)
Statistical Analysis 1: Comparison: Vibegron 75 Milligrams (mg) Once Daily (QD) vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Means Difference = -0.95, 95% CI 2-sided [-1.37 to -0.54], Standard Error of Mean 0.211

3. Secondary Outcome: Change From Baseline at Week 12 in the Average Number of Nocturia Episodes Per Night
Description: Nocturia was defined as waking to pass urine during the main sleep period. Baseline was defined as the last non-missing result on or prior to the randomization date. Change from baseline was calculated as the post-baseline value minus the baseline value.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only those participants with data available at specified time points have been presented.
Measure: Least Squares Mean (Standard Error); unit: Nocturia episodes per night
Arm/Group | Vibegron 75 Milligrams (mg) Once Daily (QD) | Placebo
Number analyzed (Participants) | 503 | 507
Nocturia episodes per night | -0.88 (0.054) | -0.66 (0.054)
Statistical Analysis 1: Comparison: Vibegron 75 Milligrams (mg) Once Daily (QD) vs Placebo; Test type: Superiority; p = 0.0015, Mixed Models Analysis; Least Squares Means Difference = -0.22, 95% CI 2-sided [-0.36 to -0.09], Standard Error of Mean 0.070

4. Secondary Outcome: Change From Baseline at Week 12 in the Average Number of Urge Urinary Incontinence (UUI) Episodes Per Day for Participants With Urinary Incontinence at Baseline
Description: The number of UUI episodes was defined as the number of times a subject checked that they had "urge" as the main reason for leakage. Average UUI episodes per day at each study visit was calculated as total number of UUI episodes within the diary analysis visit windows divided by non-missing diary days. Change from baseline was calculated as the post-baseline value minus the baseline value. Daily Averages were calculated as the sum of the event type on Complete Diary Days divided by the number of Complete Diary Days.
Time Frame: Baseline; Week 12
Population: Full Analysis Set for Incontinence (FAS-I) consists of all randomized participants with incontinence at baseline who took at least one dose of double-blind study medication, have an evaluable baseline urgency urinary incontinence measurement, and have at least one evaluable change from baseline urgency urinary incontinence measurement. Only those participants with data available at specified time points have been presented.
Measure: Least Squares Mean (Standard Error); unit: UUI Episodes Per Day
Arm/Group | Vibegron 75 Milligrams (mg) Once Daily (QD) | Placebo
Number analyzed (Participants) | 136 | 140
UUI Episodes Per Day | -2.19 (0.210) | -1.39 (0.202)
Statistical Analysis 1: Comparison: Vibegron 75 Milligrams (mg) Once Daily (QD) vs Placebo; Test type: Superiority; p = 0.0034, Mixed Models Analysis; Least Squares Means Difference = -0.80, 95% CI 2-sided [-1.33 to -0.27], Standard Error of Mean 0.269

5. Secondary Outcome: Change From Baseline at Week 12 in the International Prostate Symptom Score (IPSS) Storage Score (1-week Recall)
Description: The IPSS is based on the responses to 7 questions concerning urinary symptoms and 1 question concerning quality of life. Each question concerning urinary symptoms allows the participant to choose 1 out of 6 answers indicating increasing severity of the particular symptom. The responses are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic). Higher numerical scores represent greater severity of symptoms. Decrease in IPSS storage score indicates improvement. Baseline was defined as the last non-missing result on or prior to the randomization date. Change from baseline was calculated as the post-baseline value minus the baseline value.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only those participants with data available at specified time points have been presented.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Vibegron 75 Milligrams (mg) Once Daily (QD) | Placebo
Number analyzed (Participants) | 499 | 495
Scores on a scale | -3.0 (0.13) | -2.2 (0.13)
Statistical Analysis 1: Comparison: Vibegron 75 Milligrams (mg) Once Daily (QD) vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Means Difference = -0.9, 95% CI 2-sided [-1.2 to -0.5], Standard Error of Mean 0.17

6. Secondary Outcome: Change From Baseline at Week 12 in the Average Volume Voided Per Micturition
Description: Micturition was defined as the number of times a participant voided in the toilet as indicated on the Bladder Diary. Baseline was defined as the last non-missing result on or prior to the randomization date. Change from baseline was calculated as the post-baseline value minus the baseline value. Average volume voided per micturition at each study visit was calculated as the total volume voided over diary days within the analysis visit window divided by the total number of micturition episodes during non-missing diary days.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only those participants with data available at specified time points have been presented.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Vibegron 75 Milligrams (mg) Once Daily (QD) | Placebo
Number analyzed (Participants) | 503 | 506
mL | 25.63 (2.328) | 10.56 (2.330)
Statistical Analysis 1: Comparison: Vibegron 75 Milligrams (mg) Once Daily (QD) vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Means Difference = 15.07, 95% CI 2-sided [9.13 to 21.02], Standard Error of Mean 3.030

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: The Safety Analysis (SAS) Set includes all randomized subjects who received at least one dose of double-blind study treatment. Subjects who took any dose of Vibegron are classified as Vibegron subjects, while those who only took placebo are classified as placebo subjects. Two subjects initially randomized to placebo received Vibegron. Treatment-emergent AEs are those starting on or after the first dose of the blinded study drug, and all AE summaries cover treatment-emergent AEs in the SAS.
Arm/Group | Vibegron 75 Milligrams (mg) Once Daily (QD) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/553 | 0/551
Serious Adverse Events (participants affected / at risk) | 24/553 | 16/551
Other Adverse Events (participants affected / at risk) | 79/553 | 71/551
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibegron 75 Milligrams (mg) Once Daily (QD) (N=553) | Placebo (N=551)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bullous erysipelas (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Device lead issue (Product Issues) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Monoplegia (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative delirium (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vertebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vibegron 75 Milligrams (mg) Once Daily (QD) (N=553) | Placebo (N=551)
COVID-19 (Infections and infestations) | 22 (22) | 17 (17)
Urinary tract infection (Infections and infestations) | 14 (15) | 12 (13)
Hypertension (Vascular disorders) | 50 (53) | 46 (46)
Haematuria (Renal and urinary disorders) | 11 (11) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT03902080/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT03902080/SAP_001.pdf